CLINICAL TRIAL: NCT00991211
Title: Prospective Randomised Multicenter Study for Therapy Optimization (First Line) of Advanced Progredient, Low Malignant Non-Hodgkin Lymphomas and Mantle Cell Lymphomas
Brief Title: Bendamustine Plus Rituximab Versus CHOP Plus Rituximab
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Giessen (Other)
Responsible Party: Principal Investigator, Jurgen Barth, Study Group indolent Lymphomas (StiL), University of Giessen
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NHL 1-2003
Record Dates: First submitted 2009-10-06; First posted 2009-10-07 (Estimated); Last update posted 2024-08-22 (Actual); Status verified 2024-08

CONDITIONS: Non-Hodgkin Lymphomas; Follicular Lymphomas; Immunocytomas; Lymphocytic Lymphomas; Marginal Zone Lymphomas
Keywords: Comparison; Bendamustine + Rituximab; CHOP + Rituximab; Progression free survival; Overall survival; Toxicity; Safety
MeSH Terms: conditions — Lymphoma, Follicular; Leukemia, Lymphocytic, Chronic, B-Cell | interventions — Bendamustine Hydrochloride; Cyclophosphamide; Doxorubicin; Vincristine; Prednisone; Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Bendamustine + Rituximab (Experimental): Bendamustine 90 mg/m² d 1+2 + Rituximab 375 mg/m² d 1 q4w
  Interventions: Drug: Bendamustine
- CHOP + Rituximab (Active Comparator): Cyclophosphamid 750 mg/m² d 1 + Doxorubicin 50 mg/m² d 1 + Vincristin 1,4 mg/m² max. 2 mg d 1 + Prednison 100 mg absolute p.o. d 1-5 + Rituximab 375 mg/m² d 1 q3w
  Interventions: Drug: Standard chemotherapy CHOP + Ritiximab

INTERVENTIONS:
Drug: Bendamustine — Comparison of Bendamustine + Rituximab with CHOP + Rituximab
  Other Names: Ribomustin, Treanda
  Arms: Bendamustine + Rituximab
Drug: Standard chemotherapy CHOP + Ritiximab — Cyclophosphamid 750 mg/m² d 1 + Doxorubicin 50 mg/m² d 1 + Vincristin 1,4 mg/m² max. 2 mg d 1 + Prednison 100 mg absolute p.o. d 1-5 + Rituximab 375 mg/m² d 1 q3w as standard Chemotherapy
  Other Names: Endoxan(R), Cyclostin(R) = Cyclophosphamide; Adriamycin(R) Doxorubicin; Oncovin(R) Vincristine; Prednison; Rituxan(R), MabThera(R) = Rituximab
  Arms: CHOP + Rituximab

SUMMARY:
The study addresses the question if the first line therapy of low malignant and mantle cell lymphomas with bendamustine plus rituximab is comparable (non inferior) with CHOP plus rituximab with regard to progression free survival (PFS).

DETAILED DESCRIPTION:
The 4 agent chemotherapy (CTX) CHOP (cyclophosphamide, doxorubicin, vincristine prednisone) in combination with the monoclonal anti-CD20 antibody rituximab (CHOP-R) represents a standard CTX for the treatment of lymphomas of high or low malignancy. The combination of bendamustine and rituximab (B-R) is also highly effective with a more advantageous toxicity profile. If B-R could be shown to be non inferior to CHOP-R, this could improve the quality of life of the patient and possibly also the prognosis.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histological verified CD20-positive B-Cell-Lymphomas of the following entities:

  * Follicular lymphoma grade 1 and 2
  * Immunocytoma and lymphoplasmocytic lymphoma
  * Marginal zone lymphoma, nodal and generalised
  * Mantle cell lymphoma
  * lymphocytic lymphoma (CLL without leucaemic characteristics)
  * non-specified/classified lymphomas of low malignancy
* No prior therapy with cytotoxics,interferon or monoclonal antibodies
* Need for therapy, except mantle cell lymphomas
* Stadium III or IV
* Written informed consent
* Performance status WHO 0-2
* Histology not older than 6 months

Exclusion Criteria:

* Patients not establishing all above mentioned prerequisites
* Option of a primary, potential curative radiation therapy
* Pretreatment except a unique local delimited radiation (radiation fiel not expanding two adjacent lymph node regions
* Comorbidities excluding a study conform therapy:

  * heart attack during the last 6 months
  * severe, medicinal not adjustable hypertonia
  * severe functional defects of the heart (NYHA III or IV)
  * lung (WHO grade III or IV), liver or kidney (creatinine > 2 mg/dl, GOT + GPT or bilirubin 3 x ULN, except caused by lymphoma.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 549 (Actual)
Dates: Start 2004-01; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
Progression free survival | observation 3 years or significant differences between two arms

SECONDARY OUTCOMES:
Determination and comparison of remission rates, of toxicity, infectious complications, overall survival, EFS, TTNT, capacity of peripheral blood stem cell mobilization | ongoing

CONTACTS AND LOCATIONS:
Overall Officials: Mathias Rummel, Dr., Principal Investigator — Study Group of indolent Lymphom,as (StiL)
Locations (1):
- StiL Head Office; Justus-Liebig-University, Giessen, Germany

REFERENCES:
- [Background] Rummel MJ et al. Bendamustine Plus Rituximab Is Superior in Respect of Progression Free Survival and CR Rate When Compared to CHOP Plus Rituximab as First-Line Treatment of Patients with Advanced Follicular, Indolent, and Mantle Cell Lymphomas: Final Results of a Randomized Phase III Study of the StiL (Study Group Indolent Lymphomas, Germany). Blood 2009; 114: 405 https://doi.org/10.1182/blood.V114.22.405.405
- [Background] Rummel MJ et al. Bendamustine plus rituximab (B-R) versus CHOP plus rituximab (CHOP-R) as first-line treatment in patients with indolent and mantle cell lymphomas (MCL): Updated results from the StiL NHL 1 study. DOI: 10.1200/jco.2012.30.15_suppl.3 Journal of Clinical Oncology 30, no. 15_suppl (May 2012) 3-3.
- [Background] Rummel MJ et al. Subanalysis of the StiL NHL 1-2003 Study: Achievement of Complete Response with Bendamustine-Rituximab (B-R) and CHOP-R in the First-Line Treatment of Indolent and Mantle Cell Lymphomas Results in Superior Survival Compared to Partial Response. Blood 2012; 120: 2724.
- [Derived] Zohren F, Bruns I, Pechtel S, Schroeder T, Fenk R, Czibere A, Maschmeyer G, Kofahl-Krause D, Niederle N, Heil G, Losem C, Welslau M, Brugger W, Germing U, Kronenwett R, Barth J, Rummel MJ, Haas R, Kobbe G. Prognostic value of circulating Bcl-2/IgH levels in patients with follicular lymphoma receiving first-line immunochemotherapy. Blood. 2015 Sep 17;126(12):1407-14. doi: 10.1182/blood-2015-03-630012. Epub 2015 Aug 3. PMID 26239087
- [Derived] Rummel MJ, Niederle N, Maschmeyer G, Banat GA, von Grunhagen U, Losem C, Kofahl-Krause D, Heil G, Welslau M, Balser C, Kaiser U, Weidmann E, Durk H, Ballo H, Stauch M, Roller F, Barth J, Hoelzer D, Hinke A, Brugger W; Study group indolent Lymphomas (StiL). Bendamustine plus rituximab versus CHOP plus rituximab as first-line treatment for patients with indolent and mantle-cell lymphomas: an open-label, multicentre, randomised, phase 3 non-inferiority trial. Lancet. 2013 Apr 6;381(9873):1203-10. doi: 10.1016/S0140-6736(12)61763-2. Epub 2013 Feb 20. PMID 23433739